CLINICAL TRIAL: NCT05224726
Title: Platelet Rich Plasma for the Treatment of Uterine Scar
Brief Title: Platelet Rich Plasma for Uterine Scar
Acronym: AA-PRP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Aya Mohr Sasson, Principle investigator, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AA-PRP
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cesarean Section Complications; Uterine Bleeding; Pelvic Pain; Menstrual Irregularity
Keywords: uterine scar defect; cesarean delivery; pelvic pain; spotting; niche; cesarean section complication; uterine scar; Platelet Rich Plasma (PRP)
MeSH Terms: conditions — Uterine Hemorrhage; Pelvic Pain; Menstruation Disturbances; Metrorrhagia

STUDY DESIGN:
Intervention Model Description: Randomized control study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP Treatment (Experimental): PRP preparation will be injected to the myometrium around the uterine incision after closure of the first layer.
  Interventions: Other: Platelet Rich Plasma
- Placebo (Placebo Comparator): 0.9% of Normal Saline will be injected to the myometrium around the uterine incision after closure of the first layer.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Platelet Rich Plasma — Injection of 5cc of PRP preparation at the myometrium around the uterine incision after it has been sutured.
  Arms: PRP Treatment
Other: Placebo — Injection of 5cc of 0.9% Normal Saline at the myometrium around the uterine incision after it has been sutured.
  Arms: Placebo

SUMMARY:
When vessel wall injury occurs, platelets become activated, releasing more than 30 bioactive proteins, many of which have a fundamental role in hemostasis, inflammation and ultimate wound healing. Platelet-rich plasma (PRP), a modification of fibrin glue made from autologous blood, is being used to deliver growth factors in high concentration to sites requiring wound healing. PRP is obtained from a sample of patients' blood drawn at the time of treatment. As the rate of cesarean deliveries has been rising, long-term adverse sequelae due to uterine scar defects have been increasing. PRP might be a simple preventive treatment that potentially can reduce morbidity following cesarean deliveries.

DETAILED DESCRIPTION:
Introduction

Platelets are cytoplasmic fragments of megakaryocytes, formed in the marrow and approximately 2 μm in diameter. When vessel wall injury occurs, they become activated, releasing more than 30 bioactive proteins, many of which have a fundamental role in hemostasis, inflammation and ultimate wound healing. Growth factors released from the platelets include platelet-derived growth factor, transforming growth factor beta, platelet-derived epidermal growth factor, platelet-derived angiogenesis factor, insulin-like growth factor 1, and platelet factor 4. These factors signal the local mesenchymal and epithelial cells to migrate, divide, and increase collagen and matrix synthesis.

Platelet-rich plasma (PRP), a modification of fibrin glue made from autologous blood, is being used to deliver growth factors in high concentration to sites requiring wound healing. Its clinical uses have dramatically increased in the last decade in various fields of medicine including orthopedics, cardiothoracic surgery, plastic surgery, dermatology, dentistry, and diabetic wound healing. Recently, its positive effects in promoting endometrial and follicular growth and gestation in assisted reproduction cycles have also been demonstrated.

PRP is obtained from a sample of patients' blood drawn at the time of treatment. A 30-20 cc venous blood draw will yield 3-5 cc of PRP depending on the baseline platelet count of an individual, the device used, and the technique employed. The blood draw occurs with the addition of an anticoagulant, such as citrate dextrose to prevent platelet activation prior to its use. The preparation process requires centrifugation to separate the red blood cells (RBC) and to concentrate the platelets, which are suspended in the smallest final plasma volume. The upper 2/3 portion of the volume that is composed mostly of platelet-poor plasma (PPP) is removed. Pellets are homogenized in lower 1/3rd (5 ml of plasma) to create the Platelet-Rich Plasma (PRP). A count of 1 million /mL has become the working definition for therapeutic PRP. Activation of the platelets before their application is not required as there is no consensus for better results.

Caesarean delivery is the commonest operation performed on women worldwide with progressively rising incidence. Consequently, long-term adverse sequelae due to uterine scar defect have been increasing. Common gynecological complains include chronic pelvic pain, dyspareunia, dysmenorrhea and postmenstrual spotting and infertility. Obstetric sequelae seem to be increasing such as cesarean scar ectopic pregnancy, placenta previa, and placenta accrete, all associated with major maternal morbidity and even mortality. Given the association between uterine scar defect and gynecological symptoms, obstetric complications and potentially subfertility, it is important to develop preventive strategies.

To the best of knowledge studies using PRP for uterine scars treatment have not been published. Due to the aforementioned, the aim of our study is to learn the effect of PRP use on uterine scar healing.

Material and Methods

This is a prospective randomized double blinded study. Study population will include all women planned to undergo elective cesarean delivery at term with singleton pregnancy. Women meeting inclusion criteria will be offered to participate in the study. After signing informed consent, block randomization will be completed, including: A- administration of PRP following uterine incision repair, B - administration of placebo (0.9% normal saline) on the uterine incision. Women will be blinded to the group they have been randomized to. Blood will be drawn to all women 30 minutes before operation for platelet count and preparation of PRP (in case randomization was for group A). All operations will be performed by highly skilled surgeons of the same team. All other stages of operations will be similar in both of the groups. Operative and post-operative data will be collected from the medical files, including operation duration, estimated blood loss, operation complications (hypotension, bladder gut or vascular perforation), post-operative complications (hemorrhage, endometritis, vascular - thromboembolic event, ileus). All women will be invited to the gynecologic clinics at six weeks, 3 months and 6 months post operation for trans-vaginal sonographic evaluation of the uterine scar. Measurement will include uterine scar residual myometrial thickness (RMT), adjacent myometrial thickness (AMT), depth, length, and RMT/AMT ratio.

Women's reports regarding possibility of uterine scar defect symptoms (heavy menstrual bleeding, intermenstrual spotting, pelvic pain) will additionally be collected on follow-up visit

ELIGIBILITY:
Inclusion criteria:

* Women undergoing elective cesarean delivery
* Term pregnancy (≥37 weeks of gestation)

Exclusion criteria:

* Thrombocytopenia (CBC Platelet count <70,000)
* Connective tissue disease
* Uterine scars other than cesarean (s/p myomectomy, s/p cornual resection)
* Malformed uterus (unicornuate, bicornuate, didelphic)

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Depth of the uterine scar (mm) | At 6 weeks, 3 months, and 6 months after the cesarean delivery
  Depth of the uterine scar evaluated by transvaginal ultrasound

SECONDARY OUTCOMES:
Residual myometrial thickness/Adjacent myometrial thickness | At 6 weeks, 3 months, and 6 months after the cesarean delivery
  Ratio between adjacent and residual myometrial thickness
Niche length | At 6 weeks, 3 months, and 6 months after the cesarean delivery
  Niche length (mm)
Niche width | At 6 weeks, 3 months, and 6 months after the cesarean delivery
  Niche width evaluated by transvaginal ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Center, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dhurat R, Sukesh M. Principles and Methods of Preparation of Platelet-Rich Plasma: A Review and Author's Perspective. J Cutan Aesthet Surg. 2014 Oct-Dec;7(4):189-97. doi: 10.4103/0974-2077.150734. PMID 25722595
- [Result] Schilephake H. Bone growth factors in maxillofacial skeletal reconstruction. Int J Oral Maxillofac Surg. 2002 Oct;31(5):469-84. doi: 10.1054/ijom.2002.0244. PMID 12418561
- [Result] Sanchez AR, Sheridan PJ, Kupp LI. Is platelet-rich plasma the perfect enhancement factor? A current review. Int J Oral Maxillofac Implants. 2003 Jan-Feb;18(1):93-103. PMID 12608674
- [Result] Sharara FI, Lelea LL, Rahman S, Klebanoff JS, Moawad GN. A narrative review of platelet-rich plasma (PRP) in reproductive medicine. J Assist Reprod Genet. 2021 May;38(5):1003-1012. doi: 10.1007/s10815-021-02146-9. Epub 2021 Mar 15. PMID 33723748
- [Result] Goncalves NJN, Frantz N, de Oliveira RM. Platelet-rich plasma (PRP) therapy: An approach in reproductive medicine based on successful animal models. Anim Reprod. 2020 May 22;16(1):93-98. doi: 10.21451/1984-3143-AR2018-093. PMID 33299482
- [Result] Lin Y, Qi J, Sun Y. Platelet-Rich Plasma as a Potential New Strategy in the Endometrium Treatment in Assisted Reproductive Technology. Front Endocrinol (Lausanne). 2021 Oct 18;12:707584. doi: 10.3389/fendo.2021.707584. eCollection 2021. PMID 34733236
- [Result] Ferrari AR, Cortrezzi S, Borges E Junior, Braga D, Souza MDCB, Antunes RA. Evaluation of the Effects of Platelet-Rich Plasma on Follicular and Endometrial Growth: A Literature Review. JBRA Assist Reprod. 2021 Oct 4;25(4):601-607. doi: 10.5935/1518-0557.20210036. PMID 34415119
- [Result] Petryk N, Petryk M. Ovarian Rejuvenation Through Platelet-Rich Autologous Plasma (PRP)-a Chance to Have a Baby Without Donor Eggs, Improving the Life Quality of Women Suffering from Early Menopause Without Synthetic Hormonal Treatment. Reprod Sci. 2020 Nov;27(11):1975-1982. doi: 10.1007/s43032-020-00266-8. Epub 2020 Jul 22. PMID 32700285
- [Result] Wang CB, Chiu WW, Lee CY, Sun YL, Lin YH, Tseng CJ. Cesarean scar defect: correlation between Cesarean section number, defect size, clinical symptoms and uterine position. Ultrasound Obstet Gynecol. 2009 Jul;34(1):85-9. doi: 10.1002/uog.6405. PMID 19565535
- [Result] Tulandi T, Cohen A. Emerging Manifestations of Cesarean Scar Defect in Reproductive-aged Women. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):893-902. doi: 10.1016/j.jmig.2016.06.020. Epub 2016 Jul 5. PMID 27393285
- [Result] Semenova LS, Evlashko IuP, Sorkina NS. [Concentration of lead and several components of porphyrin metabolism in the blood and urine of persons with no industrial contact with lead]. Lab Delo. 1987;(2):11-4. No abstract available. Russian. PMID 2437359